CLINICAL TRIAL: NCT06881524
Title: A Randomized Controlled Trial of Low-Dose Amoxicillin Dual-Therapy Combined with Licorice and Lotus Root Powder for the Treatment of Helicobacter Pylori Infection
Brief Title: Low-Dose Amoxicillin Dual-Therapy Combined with Licorice and Lotus Root Powder Helicobacter Pylori Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0943
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- First-line group receiving licorice and lotus root powder combined with low-dose amoxicillin (Experimental): First-line group receiving licorice and lotus root powder combined with low-dose amoxicillin
  Interventions: Drug: First-line licorice and lotus root powder combined with low-dose amoxicillin
- First-line group receiving high-dose amoxicillin (Active Comparator)
  Interventions: Drug: First line high-dose amoxicillin
- Rescue group receiving licorice and lotus root powder combined with low-dose amoxicillin (Experimental)
  Interventions: Drug: Rescue licorice and lotus root powder combined with low-dose amoxicillin
- Rescue group receiving high-dose amoxicillin (Active Comparator)
  Interventions: Drug: Rescue high-dose amoxicillin

INTERVENTIONS:
Drug: First-line licorice and lotus root powder combined with low-dose amoxicillin — For first-line experimental group, patients would receive vonoprazan 20mg twice daily, amoxicillin 0.75g three times daily for 10 days, licorice and lotus root powder 5.0g twice daily for an additional 6 weeks
  Arms: First-line group receiving licorice and lotus root powder combined with low-dose amoxicillin
Drug: First line high-dose amoxicillin — For first-line active comparator group, patients would receive vonoprazan 20mg twice daily, amoxicillin 1 g three times daily for 10 days
  Arms: First-line group receiving high-dose amoxicillin
Drug: Rescue licorice and lotus root powder combined with low-dose amoxicillin — For rescue experimental group, patients would receive vonoprazan 20mg twice daily, amoxicillin 0.75g three times daily for 10 days, licorice and lotus root powder 5.0g twice daily for an additional 6 weeks
  Arms: Rescue group receiving licorice and lotus root powder combined with low-dose amoxicillin
Drug: Rescue high-dose amoxicillin — For rescue active comparator group, patients would receive vonoprazan 20mg twice daily, amoxicillin 1 g three times daily for 10 days
  Arms: Rescue group receiving high-dose amoxicillin

SUMMARY:
In recent years, the increasing prevalence of Helicobacter pylori (H. pylori, Hp) resistance has led to a gradual decline in the eradication rate of Hp. The growing resistance to antibiotics, particularly clarithromycin, has severely impacted the efficacy of Hp eradication. Dual-therapy regimen consisting of a proton pump inhibitor (PPI) and amoxicillin can overcome clarithromycin resistance in Hp and is effective for Hp treatment. Vonoprazan, a novel potassium-competitive acid blocker (P-CAB), has a stronger and more sustained inhibitory effect on gastric acid secretion compared to traditional PPIs. Dual-therapy regimens combining P-CABs and high-dose amoxicillin have demonstrated high eradication rates. However, the adverse effects associated with high-dose amoxicillin, such as nephrotoxicity, limit the application of this regimen. Our recent in vitro bacterial experiments and animal studies have shown that licorice, a traditional Chinese herbal medicine that is also used as a food, can inhibit the growth of Hp. This study is designed to compare a licorice-containing treatment regimen with a low-dose amoxicillin dual-therapy regimen in a clinical RCT to explore the efficacy of the former in Hp infection treatment.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori, Hp) is closely associated with chronic gastritis, peptic ulcers, gastric cancer and is classified as a Group I carcinogen. In recent years, the increasing prevalence of Hp resistance has led to a gradual decline in the eradication rate of Hp. The growing resistance to antibiotics, particularly clarithromycin, has severely impacted the efficacy of Hp eradication. Our province is considered a high-resistance area for clarithromycin and other antibiotics.

Dual-therapy regimen consisting of a proton pump inhibitor (PPI) and amoxicillin can overcome clarithromycin resistance in Hp and is effective for Hp treatment. Vonoprazan, a novel potassium-competitive acid blocker (P-CAB), has a stronger and more sustained inhibitory effect on gastric acid secretion compared to traditional PPIs. Dual-therapy regimens combining P-CABs and high-dose amoxicillin have demonstrated high eradication rates. However, the adverse effects associated with high-dose amoxicillin, such as nephrotoxicity, limit the application of this regimen.

Our recent in vitro bacterial experiments and animal studies have shown that licorice, a traditional Chinese herbal medicine that is also used as a food, can inhibit the growth of Hp. However, the role of licorice in Hp infection treatment remains to be confirmed through clinical randomized controlled trials (RCTs). Therefore, this study is designed to compare a licorice-containing treatment regimen with a low-dose amoxicillin dual-therapy regimen in a clinical RCT to explore the efficacy of the former in Hp infection treatment.

ELIGIBILITY:
Inclusion Criteria:

Age 18-70 years, regardless of sex; Positive for Helicobacter pylori (Hp); No use of proton pump inhibitors (PPIs), H2-receptor antagonists, antibiotics, or bismuth compounds within the past 4 weeks;

Exclusion Criteria:

A history of gastric or duodenal surgery; Presence of other severe comorbidities, including significant cardiac, hepatic, or renal dysfunction, malignancies, or other serious medical conditions; Allergy to any component of the investigational drug; Pregnant or breastfeeding women; Participation in another drug study within 3 months prior to enrollment in this study; Inability of the patient to accurately describe their symptoms or to comply with the requirements of this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication rate | From enrollment to the end of treatment at 6 weeks